CLINICAL TRIAL: NCT00639262
Title: Phase I Study of the Combination of Sorafenib and Radiation Therapy -/+ Temozolomide for the Treatment of Patients With Brain Metastases and Primary Brain Tumors
Brief Title: Combination of Sorafenib and Radiation for Brain Metastases and Primary Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07P.381; 2006-58 (Other: CCRRC); JT 1208 (Other: JeffTrial Number)
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases; Primary Brain Tumors
Keywords: Sorafenib; Radiation Therapy; Radiotherapy; Temozolomide; Brain Metastases; Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Sorafenib; Temozolomide; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 - Brain Metastasis (Experimental): Sorafenib and Radiotherapy
  Interventions: Drug: Sorafenib; Radiation: Radiotherapy
- Cohort 2 - Gliomas (Experimental): Sorafenib and Radiotherapy, plus Temozolomide
  Interventions: Drug: Sorafenib; Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 200mg twice daily during XRT and 30 days after. (Sorafenib will be escalated for both cohorts to determine maximum tolerated dose)
  Other Names: Nexavar
Drug: Temozolomide — For Cohort 2 - Gliomas only.
  Other Names: Temodar; Temodal
  Arms: Cohort 2 - Gliomas
Radiation: Radiotherapy — Radiation Therapy (XRT)
  Other Names: XRT; Radiation therapy; radiation oncology

SUMMARY:
Sorafenib™ has the potential to inhibit tumor growth, tumor angiogenesis , and enhance radiation response. This study will test the combination of Sorafenib™ and radiation therapy with or without temozolomide to determine tolerance of the combined treatments. Defining safe dosing of Sorafenib™ in this combination therapy will be achieved.

DETAILED DESCRIPTION:
The current standard of care for patients with brain metastatic malignancies is to receive radiation therapy alone, while the standard of care for patients with high grade primary brain malignancies, astrocytomas, is to receive to receive concurrent temozolomide with radiation therapy. In this phase I study, based on the range of efficacy of kinase inhibitors and its ability to cross the blood-brain barrier we will conduct two parallel studies. The first is to combine sorafenib and radiation therapy for the treatment of patients with brain metastases and the second is to combine sorafenib with temozolomide for primary brain tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring a minimum 2-week course of radiation therapy
2. Age > or = 18
3. All tumors of the central nervous system, or metastasis to the central nervous system.
4. Measurable disease preferred but not required for eligibility
5. Histologically or cytologically documented evidence of malignancy (for infratentorial and supratentorial glioma patients only).
6. Radiographic evidence of brain metastasis
7. ECOG performance status of 0 or 1
8. Life expectancy of > or = 3 months

Exclusion Criteria:

1. Patients receiving chemotherapy or other investigational drugs must be discontinued 14 days prior to enrollment.
2. Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
3. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
4. Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
5. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
6. Active clinically serious infection > CTCAE Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Sorafenib | 30 days post-treatment
  To determine the maximum tolerated dose (MTD) and a recommended phase II dose (RP2D) of Sorafenib and radiotherapy -/+ temozolomide patients with malignancies of the brain.

SECONDARY OUTCOMES:
Response Rate | 30 days post-treatment
  Response rate (in those patients with measurable disease)
Prediction of 1-year Recurrence | 1 year post-treatment
  Determine if an increase in urinary VEGF and MMP levels, from the end of treatment to a patient's 1-month follow-up examination, is predictive of 1-year recurrence
Safety and Toxicity of Sorafenib | 30 days post-treatment
  To evaluate the safety and toxicity profile of Sorafenib in combination with radiation therapy -/+ temozolomide

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dicker, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org